CLINICAL TRIAL: NCT06755749
Title: Effects of Family Planning (FP) Education Given to Married Illiterate Women of Reproductive Age Via Visual Material Support on FP-Related Attitudes and Contraceptive Preferences: the Case of Viranşehir
Brief Title: Effects of Family Planning Education Given to Illiterate Women Via Visual Material Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, ESRA GUNEY, PhD, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/3724
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Family Planning
Keywords: family planning; education; attitudes; contraceptive methods; midwifery
MeSH Terms: conditions — Behavior | interventions — Sex Education

STUDY DESIGN:
Intervention Model Description: randomized controlled trial conducted with experimental and control groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group receiving Family Planning Education with Visual Material Support (Experimental): Using a Family Planning Education Booklet prepared for illiterate women, an education program lasting a week in total was held in three sessions.
  Interventions: Behavioral: Family Planning Education
- Control Group (No Intervention): No intervention was made in the control group.

INTERVENTIONS:
Behavioral: Family Planning Education — Stage 1 (Day 1, 10-15 min): The education content for Session 1 in the FP Education Booklet prepared by the researchers was provided to the participants using the face-to-face interview method. After making an appointment for Stage 2 (Day 3) to be carried out at the FHC, the first stage of the data collection process was complete.
  Stage 2 (Day 3, 10-15 min): The education content for Session 2 in the FP Education Booklet was provided to the participants who arrived at the FHC on their predetermined appointment days using the face-to-face interview method. After making an appointment for Stage 3 (Day 7) to be carried out at the FHC, the second stage of the data collection process was complete.
  Stage 3 (Day 7, 1-5 min): The data collection forms were administered again to the participants who arrived at the FHC on their appointment days assigned at Stage 2, and the data collection process was complete.
  Arms: Group receiving Family Planning Education with Visual Material Support

SUMMARY:
This study was conducted to determine the effects of family planning education given to married illiterate women of reproductive age via visual material support on their family planning attitudes and contraceptive preferences.in this study, it was aimed to provide education to married illiterate women of reproductive age using visual materials to change their FP-related attitudes in a positive direction and transform these attitudes into positive fertility behaviors.

The hypotheses of the study were as follows:

H1a: FP education given with visual materials increases positive attitudes toward FP in illiterate women.

H1b: FP education given with visual materials affects the contraceptive preferences of illiterate women.

DETAILED DESCRIPTION:
This study was conducted to determine the effects of family planning education given to married illiterate women of reproductive age via visual material support on their family planning attitudes and contraceptive preferences.

Method: The randomized controlled study was carried out between 31 January and 31 July 2023. The sample of the study consisted of 148 women, including 74 in the experimental group and 74 in the control group. Using a Family Planning Education Booklet prepared for illiterate women, an education program lasting a week in total was held in three sessions. No intervention was made in the control group. Data were collected using a Personal Information Form, a Family Planning Assessment Form, and the Family Planning Attitude Scale. No intervention was made in the control group. The same data collection instruments were administered to the participants in the control group simultaneously with the experimental group in the pretest (day 1) and posttest (day 7) phases.

ELIGIBILITY:
Inclusion Criteria:

* Being able to communicate,
* Not having any visual or auditory problems that could prevent communication,
* Being aged 15-49 and married,
* Not having a diagnosis of chronic illness (e.g., cardiovascular diseases, asthma, epilepsy),
* Not receiving any FP-related education within the last 21 days.

Exclusion Criteria:

* - Being currently pregnant,
* Planning to get pregnant soon,
* Receiving medical treatment for any diagnosed chronic illness.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 74 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Family Planning Attitude | 7 days
  Its total score range is 34-170, and higher scores indicate more positive attitudes toward FP. The subscales of the scale are Attitudes of Society toward Family Planning (score range: 15-75), Attitudes of Respondent toward Family Planning (score range: 11-55), and Attitudes of Respondent toward Pregnancy (score range: 8-40).

SECONDARY OUTCOMES:
Family Planning Assessment | 7 days
  The form, which was created by the researchers by reviewing the literature, included questions about the characteristics of the participants such as the contraceptive methods they were currently using, their reasons for using (preferring) the current method, the person (self or spouse) selecting the method, previously used FP methods and reasons for quitting, the person (self or spouse) choosing to quit the method, and whether they were satisfied with the methods they used.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Güney, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared

REFERENCES:
- See also: Erenoğlu, R., & Şekerci, Y. G. (2020). Effect of training program given to the students upon family planning attitudes: a semi-experimental study. Cukurova Medical Journal, 45(3), 840-850. — https://dergipark.org.tr/en/pub/cumj/issue/54246/715555